CLINICAL TRIAL: NCT01510249
Title: A Comparison of the Analgesic Efficacies of Ultrasound and Shock Wave Therapy in the Patients With Calcaneal Spur
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Jolanta Krukowska, Head of Physical Therapy, Medical University of Lodz
Other Study IDs: JKrukowska01
Record Dates: First submitted 2011-12-16; First posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Heel Spur
Keywords: calcaneal spur; shock wave therapy; ultrasound therapy
MeSH Terms: conditions — Heel Spur

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Heel spur is a troublesome disorder. Its formation is accompanied by pain in the area of heel and it makes walking limited or even impossible.

The aim of the study is to analyze analgesic efficacy of ultrasound and shock wave therapy in patients with heel spur.

The study included 52 patients of both sexes, aged 38-86 (average 57.39) with plantar heel spur confirmed radiographically. The patients were randomly divided into two groups;in Group 1 the patients underwent ultrasound procedure (10 treatments)and in Group 2 - radial shock wave procedure(6 treatments). The researchers assessed pain three times (prior to the therapy, after the first and then the second week of treatment). In order to do this they used a modified form of the Laitinen pain indicators questionnaire (results expressed in points) and VAS - visual analogue scale (results given in milimeters). The results were statistically analyzed. In the studied periods of time a decrease in pain was observed (both in the Laitinen questionnaire and in the VAS scale). The most rapid change was noted in both the groups after the first week of treatment. Ultrasound and shock wave therapies show a comparably significant analgesic efficacy in patients with heel spur. Shock wave therapy has an advantage over ultrasound therapy. A smaller number of procedures is required to obtain comparable results, which makes the therapy less expensive. No side effects were observed during and after the treatment.

DETAILED DESCRIPTION:
The study was conducted on a group of 52 patients of both sexes, aged 38-86 years (mean 57.39; SD-11.5) with a plantar calcaneal spur confirmed by X-ray images. Patients were treated in the Department of Physical Medicine and Rehabilitation Day Unit of the University Hospital im. WAM - Central Veterans Hospital in Lodz and Municipal Health Clinic of Andrespol. In order to compare the effectiveness of the two forms of physiotherapy, ultrasound and radial shock wave therapy, the patients were randomly assigned (using a simple randomization) into two groups:

* Group 1 - ultrasound therapy group: 22 patients aged 38-86 years (mean 58.64; SD-12.99),
* Group 2 - radial shock wave group: 30 patients aged 40-71 years (mean 56.13; SD-10.02).

Ultrasound (US) was performed with a BTL 5840 S device, using labile technique, targeting the calcaneal tumor and attachment of the plantar aponeurosis (pain points); the power setting was 1,5 W/cm2, 80% fill factor, at a frequency of 1 MHz (head 4cm2). The duration of a single treatment was four minutes, and the coupling substance used was paraffin oil. Treatment sessions were performed daily Monday through Friday for a period of two weeks in a series of 10 treatments.

The shock wave therapy (SWT) was performed on the affected area using a BTL-5000 SWT device connected to a 15 mm diameter applicator according to the producer's recommendations; during therapy, 2000 strokes were applied with a frequency of 10 Hz and a capacity of 2.5 bar. Therapy took place for two weeks in a series of 6 treatments with a two-day interval between treatments.

In addition, all patients underwent kinesitherapy - exercises to strengthen the muscles that bending plantar and supinated foot to improve the mobility of the feet and to maintain the normal longitudinal arch of the foot. SPR orthopedic inserts with a pit on the painful area was used to support the longitudinal foot arch and relieve the medial ridge of the calcaneal tumor.

In all patients, pain intensity was assessed three times: before therapy, and after the first and second week of treatment. A modified form of the Laitinen indicators of pain question-shem was used [12]. On the basis of their subjective feelings, patients evaluated pain intensity, frequency of occurrence, use of analgesics, and the impact of pain on their physical activity. In addition, pain intensity was also assessed on the Huskisson visual - analogue scale (VAS) [13]; patients marked a point on a 100 mm line which corresponded to the current pain sensations - the results being given in millimeters.

The results were analyzed by Student's t-test for dependent and independent tests, with a significance level of p <0.05. The results are presented as arithmetic mean and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* plantar calcaneal spur confirmed by X-ray images

Exclusion Criteria:

* contraindications for physical therapy

Ages: 38 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted on a group of 52 patients of both sexes, aged 38-86 years (mean 57.39; SD-11.5) with a plantar calcaneal spur confirmed by X-ray images. Patients were treated in the Department of Physical Medicine and Rehabilitation Day Unit of the University Hospital im. WAM - Central Veterans Hospital in Lodz and Municipal Health Clinic of Andrespol. In order to compare the effectiveness of the two forms of physiotherapy, ultrasound and radial shock wave therapy, the patients were randomly assigned (using a simple randomization) into two groups:
  * Group 1 - ultrasound therapy group: 22 patients aged 38-86 years (mean 58.64; SD-12.99),
  * Group 2 - radial shock wave group: 30 patients aged 40-71 years (mean 56.13; SD-10.02).
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
A Comparison of the Analgesic Efficacies of Ultrasound and Shock Wave Therapy in the Patients With Calcaneal Spur | two weeks in a series of 10 ultrasound treatments and 6 radial shock wave treatments

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Krukowska, PhD, Principal Investigator — Medical University of Lodz